CLINICAL TRIAL: NCT03564496
Title: Assessment of tDCS-Induced Neuronal Responses in Multiple Sclerosis (MS) With Advanced MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-00548
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Anodal transcranial stimulation (tDCS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: Participants (N=60) (20 Healthy Controls and 40 participants with neurological disorders, ie. multiple sclerosis) will be recruited to complete self-report measures and a brief cognitive assessment and then undergo an hour long stand-alone MRI scan while simultaneously undergoing tDCS stimulation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Healthy Controls (Active Comparator): Healthy Controls will be given approximately 15 minutes of active tDCS during MRI during the initial visit.
  Interventions: Device: tDCS Administration during MRI
- MS Patients (Experimental): MS patients will be given approximately 15 minutes of active tDCS during MRI during the initial visit. After the first MRI visit, MS patients will receive remotely-supervised home tDCS treatment for a month to test the cumulative effects of tDCS. Participants will complete 20 x 2.0mA x 20 minute tDCS sessions paired with cognitive training over 4-week period (20 mins per day and weekend off) with electrodes placed to target the bilateral DLPFC. Around 3 months after the 20-session treatment, MS patients only will be asked to come to the clinic for neuropsychological assessments.
  Interventions: Device: tDCS Administration during MRI; Device: Remotely-supervised Daily tDCS Administration
- Healthy Control subgroup (Active Comparator): The Healthy Control subgroup will be given approximately 15 minutes of active tDCS during MRI during the initial visit. Participants in the healthy control subgroup will be given the option to have an additional 15 minutes of brain imaging, which will include 10 minutes of simultaneous tDCS at up to 4.0mA, added to the end of their baseline scan. After the first MRI visit, HC subgroup patients will receive remotely-supervised home tDCS treatment for a month to test the cumulative effects of tDCS. Participants will complete 20 x 2.0mA x 20 minute tDCS sessions paired with cognitive training over 4-week period (20 mins per day and weekend off) with electrodes placed to target the bilateral DLPFC.
  Interventions: Device: tDCS Administration during MRI; Device: Remotely-supervised Daily tDCS Administration; Device: Optional 15 minutes of imaging + simultaneous tDCS up to 4.0mA

INTERVENTIONS:
Device: tDCS Administration during MRI — All participants including healthy controls and MS patients will be given approximately 15 minutes of active tDCS during MRI. The simultaneous tDCS will be performed up to 2 mA dose intensity to determine CMRO2 changes from when the tDCS is on to when the tDCS is off. The stimulation consists of 15-min up to 2 mA tDCS using 5x5 cm electrode sponges with ~30s ramp-up and ramp-down periods.
Device: Remotely-supervised Daily tDCS Administration — While the first tDCS session will be performed at clinic under the full supervision, remaining sessions 2-20 (~ 1 month) will be completed at home with remote monitoring by the study technician. Participants in the HC subgroup who opt-in to the additional 15 minutes of imaging +tDCS may complete the first session remotely.
  For at-home tDCS administration, participants will be given the specially-designed tDCS device and headset, study laptop computer for secure video monitoring with study technician (must have internet access) and access to the cognitive training program, a detailed reference manual, and a training video. The device will produce up to 2.0 mA stimulation for around 20 minutes, and will not operate without the correct headset placement. The device will also automatically abort the session if optimal conditions are not maintained. It reports and records a completion code for each session.
  Arms: Healthy Control subgroup; MS Patients
Device: Optional 15 minutes of imaging + simultaneous tDCS up to 4.0mA — Participants in the healthy control subgroup who are willing may have an additional 15 minutes of imaging combined with 10 minutes of simultaneous tDCS of up to 4.0mA added at the end of their baseline scan. In this case, after the initial imaging and tDCS portion is complete, the participant will remain on the scanner for an additional 15 minutes during which brain imaging will continue and will be combined with 10 minutes of simultaneous tDCS up to 4.0mA. This will be a one-time add-on and will not be required at follow-up.
  Arms: Healthy Control subgroup

SUMMARY:
The objective of this trial is to measure the changes in neural activities during tDCS session using Magnetic Resonance Imaging (MRI). Participants (N=60) (20 Healthy Controls and 40 participants with neurological disorders, ie. multiple sclerosis) will be recruited to complete self-report measures and a brief cognitive assessment and then undergo an hour long stand-alone MRI scan while simultaneously undergoing tDCS stimulation. Methodology for this study is the administration of 15-minutes of of active tDCS during MRI acquisition compared to time without active tDCS.

ELIGIBILITY:
Inclusion Criteria for MS Patients:

* Participants must be 18 years of age or older
* Standardized SDMT Z-score > - 3.0
* Fatigue Severity Scale score > 36
* Definite MS diagnosis as assessed by licensed physician any subtype including Relapsing Remitting (RRMS), Primary Progressive (PPMS) or Secondary Progressive (SPMS)
* Score of ≤ 7.0 on the Expanded Disability Status Scale
* Clinically stable without disease progression in the past 3 months
* Has stable and continuous access to internet service at home compatible with the study laptop (Wi-Fi or Ethernet cable)
* Adequate internet capacity for remote monitoring, as tested by http://www.speedtest.net/
* Adequate home facilities (enough space, access to quiet and distraction free area)
* Able to commit to the four-week period of training sessions with baseline and two follow-up visits

Exclusion Criteria for MS Patients:

* Extreme claustrophobia
* Relapse or steroid use in previous month
* History of mental retardation, pervasive developmental disorder, or other neurological condition associated with cognitive impairment
* Primary psychiatric disorder that would influence ability to participate
* Current uncontrolled seizure disorder
* Current substance abuse disorder
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months
* Have any irremovable piercings, MRI-contraindicated implantations or metallic based-tattoos
* Pregnant or breastfeeding
* Wide Range Achievement Test-4th Edition (WRAT-4) Reading Recognition Scaled Score < 85
* Beck Depression Inventory - Fast Screen (BDI-FS) score > 9

Inclusion Criteria for Healthy Controls:

* Participants must be 18 years of age or older
* Standardized SDMT Z-score > - 3.0
* Have not been diagnosed with MS or other neurological disorder
* Adequate internet capacity for remote monitoring, as tested by http://www.speedtest.net/ (HC subgroup only)
* Adequate home facilities including enough space, access to quiet and distraction free area (HC subgroup only)
* Able to commit to the four-week period of training sessions with baseline and one follow-up visit (HC subgroup only)

Exclusion Criteria for Healthy Controls:

* Extreme claustrophobia
* History of mental retardation, pervasive developmental disorder or other neurological condition associated with cognitive impairment
* Primary psychiatric disorder that would influence ability to participate
* Current uncontrolled seizure disorder
* Current substance abuse disorder
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months
* Have any irremovable piercings, MRI-contraindicated implantations or metallic based-tattoos
* Pregnant or breastfeeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data collection will be for pilot data and exploratory analysis.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | MS Patients | Healthy Control Subgroup
Started | 27 | 40 | 6
Completed | 26 | 36 | 6
Not Completed | 1 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Screen failure | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | MS Patients | Healthy Control Subgroup | Total
Number analyzed (Participants) | 26 | 36 | 6 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (15.8) | 47 (14.7) | 36 (14.54) | 39.6 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 3 | 41
  Male | 11 | 13 | 3 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 23 | 32 | 5 | 60
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 0 | 11
  White | 10 | 23 | 5 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 0 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 36 | 6 | 68

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Metabolic Rate of Oxygen (CMRO2)
Description: Measured via MRI. CMRO2 is the amount of O2 the brain consumes per unit of time (in μmol O2/100g tissue per minute)
Time Frame: Baseline Visit
Measure: Mean (Standard Deviation); unit: µmol/100g/min
Arm/Group | Healthy Controls | MS Patients | Healthy Control Subgroup
Number analyzed (Participants) | 23 | 20 | 6
µmol/100g/min | 165.84 (25.32) | 128.3 (14) | 159.4 (21.8)

2. Primary Outcome: Cerebral Metabolic Rate of Oxygen (CMRO2)
Description: Measured via MRI. CMRO2 is the amount of O2 the brain consumes per unit of time (in μmol O2/100g tissue per minute)
Time Frame: Intermediate Visit (Month 1)
Population: Only the Healthy Control subgroup and MS patients were evaluated for this outcome measure. The Healthy Control group was not evaluated because they did not receive any additional sessions after the first visit.
Measure: Mean (Standard Deviation); unit: µmol/100g/min
Arm/Group | Healthy Control Subgroup | MS Patients
Number analyzed (Participants) | 5 | 20
µmol/100g/min | 146.42 (27.71) | 140.59 (13.83)

3. Primary Outcome: Neuronal Reactivity (NR)
Description: NR represents tDCS-induced global neural reactivity measured by CMRO2 levels in cells available to respond to neural stimuli. NR is measured as the percentage change of CMRO2 from no tDCS to real tDCS. tDCS will be administered in one visit and will last for approximately 15 minutes.
Time Frame: Baseline Visit (pre-tDCS, post-tDCS)
Measure: Mean (Standard Deviation); unit: percentage change of CMRO2
Arm/Group | Healthy Controls | MS Patients | Healthy Control Subgroup
Number analyzed (Participants) | 23 | 20 | 5
percentage change of CMRO2 | 9.84 (10.8) | 12.45 (13.8) | 15.61 (4.69)

4. Primary Outcome: Neuronal Reactivity (NR)
Description: NR represents tDCS-induced global neural reactivity measured by CMRO2 levels in cells available to respond to neural stimuli. NR is measured as the percentage change of CMRO2 from no tDCS to real tDCS.
Time Frame: Baseline, Intermediate Visit (Month 1)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change of CMRO2
Arm/Group | MS Patients | Healthy Control Subgroup
Number analyzed (Participants) | 20 | 5
percentage change of CMRO2 | 4.32 (8.44) | 22.5 (6.88)

5. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QOL) Score
Description: 36-item assessment of quality of life measures in participants with neurological disorders. This questionnaire will be administered to MS patients only. The raw score is the sum of responses; this score is transformed to a standardized T-score with a mean of 50 and SD of 10. A T-score of 60 indicates worse (undesirable) self-reported health.
Time Frame: Baseline Visit
Population: Only MS patients were evaluated for this outcome measure. The Healthy Control group and Health Control subgroup were not administered the Neuro-QOL.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- MS Patients: Individuals diagnosed with MS recruited from the MS Center/ Neurology Department at NYULMC
  Active tDCS: The simultaneous tDCS will be performed at up to 2 mA dose intensity to determine CMRO2 changes from when the tDCS is on when the tDCS is off. The stimulation (left anodal at DLPFC regions) consists of 15-min up to 4 mA tDCS using 5x5 cm electrode sponge with ~30s ramp-up and ramp-down periods.
  Sham (placebo) stimulation: MRI-compatible tDCS off (immediately before and after tDCS)
Arm/Group | MS Patients
Number analyzed (Participants) | 31
T-score | 50.81 (13.04)

6. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QOL) Score
Description: as for outcome 5
Time Frame: Intermediate Visit (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MS Patients
Number analyzed (Participants) | 26
T-score | 36.38 (13.16)

7. Secondary Outcome: Quality of Life in Neurological Disorders (Neuro-QOL) Score
Description: as for outcome 5
Time Frame: Final Visit (Month 4)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MS Patients
Number analyzed (Participants) | 29
T-score | 39.12 (12.65)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Systematic assessment through self-reported questionnaires.
Arm/Group | Healthy Controls | MS Patients | Healthy Control Subgroup
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/36 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/36 | 0/6
Other Adverse Events (participants affected / at risk) | 20/26 | 27/36 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Controls (N=26) | MS Patients (N=36) | Healthy Control Subgroup (N=6)
Tingling (Skin and subcutaneous tissue disorders) | 8 | 14 | 0
Itching (Skin and subcutaneous tissue disorders) | 6 | 4 | 0
Warmth Sensation under the electrode (Skin and subcutaneous tissue disorders) | 6 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT03564496/Prot_SAP_000.pdf